CLINICAL TRIAL: NCT05253677
Title: Precise Procedural and PCI Plan (P4) Randomized Clinical Trial Integration of Coronary Computed Tomography Angiography in the Catheterization Laboratory to Plan and Guide Coronary Percutaneous Procedures
Brief Title: Precise Procedural and PCI Plan (P4)
Acronym: P4
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CoreAalst BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRI-052
Record Dates: First submitted 2021-12-06; First posted 2022-02-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-guided PCI strategy (Experimental): QAngio CT Research Edition is a software suite providing several functionalities for the analysis of coronary computed tomography angiography (CCTA) scans to extract and present relevant information on the coronary vasculature for further clinical investigation.
  Also, QAngio CT Research Edition allows to export this information for later viewing during x-ray angiography (XA) procedures to help physicians plan and guide the interventional procedure.
  Interventions: Device: CT-guided PCI
- intravascular ultrasound (IVUS)-guided PCI strategy (Active Comparator): Intravascular ultrasound (IVUS) is an invasive intravascular imaging technique able to visualize the coronary vessel. The use of IVUS-guided PCI has been endorsed an recommended by the European Society of Cardiology. The device is considered part of standard of clinical care.
  Interventions: Device: IVUS-guided PCI

INTERVENTIONS:
Device: CT-guided PCI — CT-guided PCI with standardized pre-procedural planning and online guidance.
  Arms: CT-guided PCI strategy
Device: IVUS-guided PCI — use of IVUS during PCI procedure (standard of care)
  Arms: intravascular ultrasound (IVUS)-guided PCI strategy

SUMMARY:
Computed tomography (CT) has become an established tool in the diagnostic workup of patients with suspected coronary artery disease (CAD). The availability of coronary CT angiography (CCTA) before the invasive procedure allows stratifying case complexity and can be used to improve patient selection for PCI, to plan and guide therapeutic interventions. Beyond the diagnostic and therapeutic phase, it helps to better organize the catheterization laboratory workflow.

The P4 study is an investigator-initiated, multicenter, randomized study with a non-inferiority design of patients with an indication for PCI aiming at comparing clinical outcomes between two imaging strategies to guide PCI, being coronary CT-guided PCI strategy (investigational technology) and IVUS-guided PCI strategy (comparator).

After identifying the presence of a significant coronary stenosis, the patient will be randomized either to CT- or IVUS-guided PCI groups. Both CT and IVUS-guided PCI will be performed following the P4 trial protocol. When the procedure is completed, post-PCI FFR will be measured. All patients will be followed in hospital, at 30 days (±15 days), 12 months (±1 month) and yearly until 5 year.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be at least 18 years of age and younger than 80 years old.
2. Subject must have evidence of myocardial ischemia (e.g., stable angina, silent ischemia (ischemia in the absence of chest pain or other anginal equivalents), unstable angina, or acute myocardial infarction) suitable for elective PCI.
3. Patients with a clinical indication for revascularization presenting with stable coronary artery disease or stabilized acute coronary syndrome defined as follows unstable angina (Braunwald class IB, IC, IIB, IIC, IIIB, IIIC), patients with NSTEMI without high-risk features such as recurrence of chest pain, ST-segment depression>1mm in ≥6 leads plus ST-segment elevation in aVR, life-threatening arrhythmias, mechanical complications of MI, resuscitated cardiac arrest, GRACE risk score>140.
4. All target lesions must be planned for treatment only in vessels with RVD ≥2.5 mm and ≤4.0 mm.
5. No more than 2 target vessels are allowed. A bifurcation counts as a single lesion even if the side branch is planned to be treated.
6. Subject must provide written Informed Consent before any study-related procedure.

Exclusion Criteria:

1. Age <18 years or ≥80 years old
2. STEMI as clinical presentation.
3. Uncontrolled or recurrent ventricular tachycardia.
4. Hemodynamic instability.
5. Severe renal dysfunction, defined as an eGFR ≤30 mL/min/1.73 m2.
6. Atrial fibrillation, flutter, or arrhythmias.
7. Previous PCI or CABG.
8. The target lesion is in the left main coronary artery
9. BMI ≥35 kg/m2.
10. Insufficient CT quality assessed by the Core lab.
11. Comorbidity with life expectancy ≤ 2 years.
12. Inability to take DAPT (both aspirin and a P2Y12 inhibitor) for at least 12 months in the patient presenting with an ACS, or at least 6 months in the patient presenting with stable CAD, unless the patient is also taking chronic oral anticoagulation in which case a shorter duration of DAPT may be prescribed per local standard of care.
13. Planned major cardiac or non-cardiac surgery within 24 months after the index procedure Note: Major surgery is any invasive operative procedure in which an extensive resection is performed, e.g., a body cavity is entered, organs are removed, or normal anatomy is altered. Note: Minor surgery is an operation on the superficial structures of the body or a manipulative procedure that does not involve a serious risk. Planned minor surgery is not excluded.
14. Prior PCI within the target vessel within 12 months.
15. Subject has known hypersensitivity or contraindication to any of the study drugs (including all P2Y12 inhibitors, one or more components of the study devices, including everolimus, zotarolimus, biolimus, sirolimus, cobalt, chromium, nickel, platinum, tungsten, acrylic, and fluoropolymers, or radiocontrast dye that cannot be adequately pre-medicated.
16. The subject has received a solid organ transplant that is functioning or is active on a waiting list for any solid organ transplants with expected transplantation within 24 months.
17. The subject receives immunosuppressant therapy or has known immunosuppressive or severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.). Note: corticosteroids are not included as immunosuppressant therapy.
18. The subject has previously received or is scheduled to receive radiotherapy to a coronary artery (vascular brachytherapy) or the chest/mediastinum.
19. Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
20. The subject has a documented or suspected hepatic disorder as defined as cirrhosis or Child-Pugh ≥ Class B.
21. The subject has a history of bleeding diathesis or coagulopathy or has had a significant gastro-intestinal or significant urinary bleed within the past six months. The subject has had a cerebrovascular accident or transient ischemic neurological attack (TIA) within the past six months, or any prior intracranial bleed, or any permanent neurologic defect, or any known intracranial pathology (e.g., aneurysm, arteriovenous malformation, etc. The subject has a life expectancy <2 years for any non-cardiac cause.
22. Subject is currently participating in another investigational drug or device clinical study.
23. Pregnant or nursing subjects and those who plan pregnancy in the period up to 2 years following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.
24. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
25. Unable to provide written informed consent (IC).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1090 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
rate of MACE between CCTA- and IVUS-guided PCI strategy | 12 months follow-up
  Comparison of the rate of the composite of major adverse cardiovascular events, defined as cardiac death, target vessel myocardial infarction, and ischemia-driven target vessel revascularization between CT- and IVUS-guided PCI strategies at 12-month follow-up

SECONDARY OUTCOMES:
Compare in-hospital resource utilization between CCTA- and IVUS-guided PCI strategies. | during the intervention
  Compare in-hospital resource utilization (cost from all the procedures during the hospitalisation to discharge in Euros) between CCTA- and IVUS-guided PCI strategies.
Compare resource utilization at 12-month follow-up between CCTA- and IVUS-guided PCI strategies | 12 months follow-up
  Compare resource utilization (procedural cost and cost from additional interventions in Euros) at 12-month follow-up between CCTA- and IVUS-guided PCI
Compare radiation dose (defined as radiation dose from the invasive procedure) between CCTA- and IVUS- guided PCI strategies. | periprocedural time frame
Compare contrast volume (defined as contrast volume used during the invasive procedure) between CCTA- and IVUS- guided PCI strategies. | periprocedural time frame
Compare the rate of cardiac death between CCTA- and IVUS-guided PCI strategies. | 12 months follow-up
Compare the rate of target-vessel myocardial infarction between CCTA- and IVUS-guided PCI strategies. | 12 months follow-up
Compare the rate of ischemia-driven target-vessel revascularization between CCTA- and IVUS-guided PCI strategies. | 12 months follow-up
Compare the rate of PCI-related MI (type 4a a, 4th Universal Definition of MI) between CCTA- and IVUS-guided PCI strategies | during the procedure
Compare the degree of functional revascularization, defined by post-PCI FFR values measured immediately after PCI between CCTA- and IVUS-guided PCI strategies. | periprocedural time frame
Compare the degree of functional revascularization, defined by FFRCT Planner, between CCTA- and IVUS-guided PCI strategies. | periprocedural time frame
Compare the rate of MACE between patient with complete and incomplete functional revascularization based on the FFRCT Planner, at 12-month follow-up. | 12 months follow-up
Compare the rate of MACE between patient with complete and incomplete functional revascularization based on the post-PCI FFR values measured immediately after PCI, at 12-month follow-up. | 12 months follow-up
Assess the agreement on post-PCI FFR between the FFRCT Planner and the invasive measurement. | periprocedural time frame
Assess the agreement between the FFRCT Planner strategy and the actual treatment performed. | periprocedural time frame
Assess the CCTA predictors of stent under expansion. | periprocedural time frame
  To assess which characteristics of the plaque, defined by CT, can predict whether the stent is under expansion (by multivariate analysis on the data)
To compare angiographic Endpoints (Core Lab assessed QCA): - Final (post-PCI) minimal lumen diameter. - Final (post-PCI) percent diameter stenosis. - Acute lumen gain post-intervention. | periprocedural time frame
To compare the maximum device size (stent or post-dilatation balloon)/reference vessel diameter ratio) CCTA- and IVUS-guided PCI strategies. | periprocedural time frame
To compare angiographic complications CCTA- and IVUS guided PCI strategies. | periprocedural time frame
  Angiographic dissection ≥ NHLBI type B, perforations (Ellis's classification), intra-procedural thrombotic events (including slow-flow, no-reflow, side branch closure, distal embolization, and intra-procedural stent thrombosis, as per the standard angiographic core laboratory definitions
To compare procedural time (defined as the time from first to the last angiography) between CCTA- and IVUS-guided PCI strategies. | periprocedural time frame
Compare the rate of symptoms-free status assessed by the SAQ-7 between CCTA- and IVUS-guided PCI strategies at 12-months. | 12 months follow-up
Compare the change in symptoms assessed by the change of Seattle Angina Questionnaire (SAQ-7) scores between CCTA- and IVUS-guided PCI strategies at 12-months. | 12 months follow-up
Compare the change in symptoms assessed by the change of EuroQol 5 dimensions - 5 levels (EQ-5D-5L) scores between CCTA- and IVUS-guided PCI strategies at 12-months. | 12 months follow-up
Assess the capacity of the FFRCT Planner (predicted post-PCI FFR) to predict adverse events. | 12 months follow-up
  Assess whether the predicted post-PCI FFR value which is calculated by the FFRCT-planner can predict adverse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Collet Bortone, MD, PhD, Principal Investigator — CoreAalst BV; Daniele Andreini, MD, PhD, Principal Investigator — Milan University, Milan, Italy
Locations (23):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - St. Francis Hospital & Heart Center, Roslyn, New York
- Belgium (3):
  - UZ Brussels, Jette, Brussels Capital
  - OLV Hospital, Aalst
  - Hartcentrum ZNA Antwerp, Antwerp
- Denmark (3):
  - Gentofte hospital, Gentofte Municipality, Hellerup
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet, Copenhagen
- Centre Hospitalier Universitaire de Lille, Lille, France
- Medical Imaging Centre, Semmelweis University, Budapest, Hungary
- Italy (4):
  - Azienda Ospedaliero Universitaria di Ferrara, Cona
  - Humanitas University, Milan
  - Ospedale Galeazzi Sant'Ambrogio, Milan
  - Centro Cardiologico Monzino S.P.A., Milan
- Aichi Medical University, Aichi, Japan
- United Kingdom (7):
  - University Hospitals Dorset NHS Foundation Trust, Poole Hospital, Poole, Dorset
  - Golden Jubilee National Hospital, Clydebank
  - Liverpool Heart and Chest Hospital, Liverpool
  - St George's University Hospitals NHS Foundation Trust, London
  - Barts Health NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Freeman Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: No